CLINICAL TRIAL: NCT06615453
Title: A Prospective Study Assessing the Impact of Tixel Treatment of Peri Orbital Wrinkles on Symptoms and Signs in Patients With Dry Eye Disease
Brief Title: Impact of Tixel Treatment on Symptoms and Signs in Patients With Dry Eye Disease
Acronym: TIXEL-DED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLS21162; RECID HLS21162 (Other: Aston University)
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry eye disese, Tixel treatment
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tixel treatment (Experimental)
  Interventions: Device: Thermo-mechanical action based peri-orbital fractional skin treatment
- Sham treatment (Sham Comparator)
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Thermo-mechanical action based peri-orbital fractional skin treatment — Participants will receive three Tixel® treatments at 2-weeks intervals
  Arms: Tixel treatment
Device: Sham treatment — Participants will receive three sham treatments at 2-weeks intervals
  Arms: Sham treatment

SUMMARY:
This study will examine how a standard Tixel treatment versus a sham treatment for eye wrinkles affects the symptoms and signs of Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to Moderate Periorbital wrinkles
2. OSDI score of at least 23
3. Noninvasive Tear film break up time (NIBUT) ≤ 10 seconds
4. No other eye or skin or immune problems
5. Willing and able to provide written informed consent.
6. Willing to participate in all study activities and instructions.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding
2. Lesions in the periorbital area
3. Acute severe blepharitis
4. Acute conjunctivitis
5. Use of eye drops within 2 hours before examination
6. Other concomitant anterior eye disease
7. Has undergone outdoors/sunbed tanning during the last 4 weeks
8. Is unwilling to follow the Tixel aftercare instructions after each of the three Tixel treatments.
9. Active Herpes Simplex or tendency for Herpes Simplex in the periorbital area (meaning the subject has had the condition previously).
10. Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
11. An impaired immune system condition or use of immunosuppressive medication.
12. Collagen disorders, keloid formation and/or abnormal wound healing.
13. Previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans for such treatment during the course of the Tixel2 device treatment, or before complete healing of such treatments has occurred.
14. Any patient who takes or has taken any medications (including via topical application), herbal treatment (oral or topic), food supplements or vitamins, which may cause fragile skin or impaired skin healing during the last 3 months.
15. Any patient who has used oral Isotretinoin (Accutane® or Roaccutan®) within 3 months prior to treatment or less.
16. Any patient who has a history of bleeding coagulopathies or use of anticoagulants.
17. Any patient who has tattoos or permanent makeup in the treated area.
18. Any patient who has burned skin, blistered skin, irritated skin, or sensitive skin in any of the areas to be treated.
19. Any patient who underwent thread lifting of the area to be treated in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of periorbital Tixel treatments in patients with dry eye through the reporting of adverse events (AE) and serious adverse events (SAE) exclusively. | Through study completion, an average of 4 months
  SAFETY, number of AEs Any safety related event during the study will be recorded and analyzed

SECONDARY OUTCOMES:
To evaluate the impact of the treatment on symptoms and signs of dry eyes and compare the findings with those of a control group. | Through study completion, an average of 4 months
  NIBUT Seconds OSDI Score Topography mm/ D Slit Lamp examination Standardized Patient Evaluation of Eye Dryness (SPEED) Questionnaire Lid margin profile Tear Sampling Analysis Ocular tear biomarkers Meibography Corneal staining with fluorescein Conjunctival staining with lissamine green

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Science, School of Optometry, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided